CLINICAL TRIAL: NCT06625645
Title: Comparative Evaluation of Antimicrobial Efficacy, Clinical and Radiographic Success of Calcium Hydroxide, Chlorhexidine, and Modified Triple Antibiotic Paste in Different Combination Forms As Intracanal Medicaments Against Enterococcus Faecalis in Primary Teeth: a Randomized Clinical Trial
Brief Title: Comparative Evaluation of Antimicrobial Efficacy, Clinical and Radiographic Success of Calcium Hydroxide, Chlorhexidine, and Modified Triple Antibiotic Paste in Different Combination Forms As Intracanal Medicaments Against Enterococcus Faecalis in Primary Teeth
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mahy Abdel Raouf Aly Kamar (Other)
Responsible Party: Sponsor-Investigator, Mahy Abdel Raouf Aly Kamar, Principle investigator, Cairo University
Organization: Cairo University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 14422023573623; main investigator (Registry Identifier: Mahy Abdel Raouf)
Record Dates: First submitted 2024-09-28; First posted 2024-10-03 (Actual); Last update posted 2024-10-17 (Actual); Status verified 2024-10

CONDITIONS: Apical Periodontitis; Necrotic Primary Molars; Periapical Pathosis of Primary Molars
Keywords: Necrotic Primary Teeth; Apical Periodontitis; Non Vital primary teeth; periapical pathosis of primary teeth; intracanal medication; triple antibiotic paste; enterococcus faecalis; Microbiology; bacterial reduction
MeSH Terms: conditions — Periapical Periodontitis | interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Calcium Hydroxide mixed with saline as control intracanal medication (Active Comparator): using calcium hydroxide with saline as control intracanal medication for necrotic primary molars
  Interventions: Combination Product: calcium hydroxide mixed with saline as intracanal medication
- different types and combinations of intracanal medications for necrotic primary molars (Experimental)
  Interventions: Combination Product: Modified triple antibiotic paste (TAP) mixed with chlorehexidine; Combination Product: Modified Triple Antibiotic Paste mixed with saline; Combination Product: Calcium Hydroxide mixed with chlorohexidine Intracanal medication

INTERVENTIONS:
Combination Product: Modified triple antibiotic paste (TAP) mixed with chlorehexidine — M-TAP with CHX 2%
  Arms: different types and combinations of intracanal medications for necrotic primary molars
Combination Product: Modified Triple Antibiotic Paste mixed with saline — M-TAP mixed with saline
  Arms: different types and combinations of intracanal medications for necrotic primary molars
Combination Product: Calcium Hydroxide mixed with chlorohexidine Intracanal medication — calcium hydroxide powder mixed with CHX 2% solution as intracanal medication
  Arms: different types and combinations of intracanal medications for necrotic primary molars
Combination Product: calcium hydroxide mixed with saline as intracanal medication — calcium hydroxide mixed with saline as intracanal medication for necrotic primary molars
  Arms: Calcium Hydroxide mixed with saline as control intracanal medication

SUMMARY:
Comparing between different intracanal medications with different combination forms of Modified Triple Antibiotic Paste, Calcium Hydroxide and Chlorehexidine, regarding antimicrobial efficacy through bacterial reduction count of enterococcus Faecalis and regarding clinical and radiographic success in non vital primary teeth necessitating pulpectomy with follow up time 1 year.

DETAILED DESCRIPTION:
1. Full medical and dental history will be obtained from the parents of the patients participating in this study.
2. A thorough clinical and radiographic examination of the tooth to be treated will be done.
3. The tooth will be anaesthetized using the inferior alveolar nerve block technique for lower molars and infiltration for upper molars
4. Before isolation, antisepsis of the oral cavity will be performed by rinsing for 1 min with 10 mL chlorhexidine gluconate mouth-wash 0.2 %.
5. The tooth will be properly isolated using rubber dam.
6. Access cavity will be performed using a round bur.
7. The root canals will be irrigated with 1 ml sterile saline solution.
8. Patency of the root canal will be obtained using stainless steel hand k- files size #15
9. Working length will be determined using apex locator
10. The first microbial samples (S1) will be collected to assess bacterial count of the root canals using 1 sterile paper point size 20, which will be inserted into the widest root canal for 1 min with pumping movements (McGurkin-Smith et al., 2005)
11. It will be placed inside sterile tubes containing a reduced transport medium of thioglycolate.
12. The canals will be thoroughly irrigated using 3ml syringe of 1.25% Sodium hypochlorite. A side-vented needle will be used to control the possibility of irrigant apical extrusion.
13. Mechanical preparation will be performed with rotary system for all the cases.
14. Irrigation with saline solution will be used to neutralize all the previously used solutions.
15. Then, a second microbial samples (S2) representing the antibacterial effect of the mechanical preparation will be obtained with the same procedure as the first sample (S1).
16. According to the randomization sequence, patients will be assigned to one of 4 groups:

1- A mix of modified triple Antibiotic Paste (M-TAP) and normal saline (experimental).

2- A mix of Ca(OH)2 and 2% CHX gluconate solution(experimental). 3- A mix of M-TAP and 2% CHX gluconate solution(experimental). 4- A mix of Ca(OH)2 and normal saline (control) 17) The canals will be dried and filled with intracanal medication plugged into the canal by using a plugger.

18) At the end of the first visit a piece of sterile cotton will be placed in the pulp chamber.

19) All teeth will be dressed with intermediate restorative material (IRM) as a temporary filling, in order to ensure proper sealing with no leakage of any oral fluids inside the root canal, which might disturb the action of the intracanal medication.

20) After 7 days, the temporary restoration will be removed. 21) Disinfection of the operative field will take place as performed previously using the same protocol.

22) Irrigation of the root canals with 2 mL of saline to flush out the medicaments and the third bacteriological sample (S3) will be taken out.

23) Later, canals will be filled with Metapex (Metabiomed, Korea), followed by the placement of stainless-steel crowns (3M ESPE).

24) The samples will be placed in sterile vials with thioglycolate (transport medium). The vials will be sealed tightly to avoid contamination and labeled. The labeled vials will be kept in a freezer and will be sent to the laboratory within 1 hour of collection, and samples will be assessed for total E. faecalis count (Qamar et al., 2023).

ELIGIBILITY:
Inclusion Criteria:

• Primary molars necessitating pulpectomy diagnosed with deep dental caries with pulp necrosis, apical periodontitis and periapical pathosis or both.

* Non-Vital pulps.
* Negative response to hot or cold pulp tester (ethyl chloride spray ).
* Decayed tooth with spontaneous unprovoked long dull aching pain showing signs of necrosis of the pulp

Exclusion Criteria:

* Medically compromised and uncooperative children
* Tooth indicated for extraction
* Mobile teeth (Miller's Grade 2 or more)
* teeth with more than two-thirds of root resorption
* previous endodontic treatment

Ages: 4 Years to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 32 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2025-05-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Enterococcus faecalis bacterial reduction | 3 times, one after the access and gaining patency, second one after chemomechanical preparation and the third one after 7 days from intracanal medication insertion in the canal
  Samples from canal using paper point size 20 with pumping action from the widest canal three times one after the access and gaining patency, second one after chemomechanical preparation and the third one after 7 days from intracanal medication insertion in the canal, then the samples will be placed in sterile vials with thioglycolate (transport medium). The vials will be sealed tightly to avoid contamination and labeled. The labeled vials will be kept in a freezer and will be sent to the laboratory within 1 hour of collection, and samples will be assessed for total E. faecalis count.

SECONDARY OUTCOMES:
Clinical success | 3,6 and 12 months
  measuring pain through presence or absence of pain Visual inspection of any changes (Redness or swelling of vestibular area (presence or absence of any change) Tenderness upon percussion ( positive or negative response) Tenderness upon touching of the vestibulum ( positive or negative response)

OTHER OUTCOMES:
Radiographic success | 6 and 12 months
  Digital periapical radiographs for assessing the integrity of the pulp and surrounding structures.
  Periodontal ligament (PDL) widening, loss of lamina dura, internal or external root resorption, and radiolucency of furcation or periapical pathosis) will be considered as a failure with dichotomous response (yes/no)

IPD SHARING:
Plan to Share IPD: No